CLINICAL TRIAL: NCT06220006
Title: Lesion Formation With Pulsed Field Versus Cryobaloon Ablation as Assessed by Cardiac Magnetic Resoncance
Acronym: PULSED-ICE-CMR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Ivo Roca, Head of Arrhythmia Section. Professor of Cardiology, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PULSED-ICE-CMR
Record Dates: First submitted 2023-09-18; First posted 2024-01-23 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Catheter ablation; Ablation lesion; Pulmonary vein isolation; Pulsed field ablation; Cryoballoon ablation; Cardiac magnetic resonance; Late gadolinium enhancement
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pulsed Field Ablation (Experimental): Pulmonary vein isolation using the Farapulse Pulsed Field Ablation System (Boston Scientific)
  Interventions: Procedure: Pulmonary vein isolation
- Cryoballoon Ablation (Active Comparator): Pulmonary vein isolation using the Medtronic Cryoballoon Ablation System
  Interventions: Procedure: Pulmonary vein isolation

INTERVENTIONS:
Procedure: Pulmonary vein isolation — Catheter ablation

SUMMARY:
This randomised study will compare pulsed field ablation and cryoballoon ablation with respect to ablation lesion quality as assessed by late gadolinium enhancement (LGE) cardiac magnetic resonance (CMR) at 3 months post-ablation. Patients scheduled for first-time AF ablation will be randomised in a 2:1 fashion to receive PVI-only, either by pulsed field ablation (Farapulse Pulsed Field Ablation System, Boston Scientific) or cryoballoon ablation (Medtronic Cryoballoon Ablation System).

DETAILED DESCRIPTION:
Pulmonary vein isolation (PVI) using catheter ablation has become a cornerstone in the treatment of AF and is considered the most effective therapy today. Catheter ablation has been mostly performed employing thermal energies, with radiofrequency and cryo-balloon ablation being the best validated most widely applied modalities. Despite substantial technological and procedural advances that have improved efficacy, efficiency and safety of AF ablation in recent years, long-term durability of ablation lesions is still not satisfactory, and rare but potentially life-threatening procedure-related complications like cardiac tamponade or atrio-esophageal fistula remain a concern. In addition, phrenic nerve palsy complicates a relevant proportion of procedures, particularly in cryo-ablation.

The novel non-thermal ablation method of pulsed field ablation holds great promise in that respect. Pulsed field ablation achieves permanent cell death through electroporation, which appears to provide a unique selectivity for cardiomyocytes and to spare surrounding tissues composed of other cell types, thus minimising the risk of collateral damage.This method has already been introduced into routine clinical practice and is established in many centers worldwide. A large number of studies have confirmed safety and efficacy of pulsed field ablation for pulmonary vein isolation in the context of AF and found significant reductions in ablation times. However, the putative benefits regarding efficacy, efficiency and safety remain to be proven in randomised controlled trials.

Against this background, the investigators aim to perform a randomised clinical trial comparing pulsed field ablation with thermal cryo-balloon ablation with respect to efficacy, effectiveness and safety. Patients scheduled for first-time AF ablation will be randomised in a 2:1 fashion to receive PVI-only, either by pulsed field ablation (Farapulse Pulsed Field Ablation System, Boston Scientific) or cryoballoon ablation (Medtronic Cryoballoon Ablation System). The primary outcome of this trial will be ablation lesion quality as assessed by late gadolinium enhancement (LGE) cardiac magnetic resonance (CMR) at 3 months post-ablation.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for first-time atrial fibrillation catheter ablation

Exclusion Criteria:

* age <18 years
* long-standing persistent atrial fibrillation
* prior left atrial ablation
* pregnancy or lactation
* reduced left ventricular ejection fraction
* GFR <30%
* BMI >35%
* left atrial diameter >55 mm
* cardiac implantable electronic device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
LGE-CMR-determined ablation lesion quality | 3 months post-ablation
  Complete late gadolinium enhancement encircling both pulmonarz vein pairs, with discontinuations adding up to less than 10% of the total length of the circumference

SECONDARY OUTCOMES:
AF-free survival | 3, 6 and 12 months post-ablation
Arrhythmia-free survival | 3, 6 and 12 months post-ablation
  Freedom from atrial tachycardia, atrial flutter and AF
Time to first AF recurrence | 12, 24 and 36 months
Progression from paroxysmal to persistent AF | 12, 24 and 36 months
Time to first arrhythmia | 12, 24 and 36 months
Spatial LGE distribution according to local wall thickness (as assessed by preablation CT) | 3 months post-ablation
Complete pulmonary vein isolation confirmed by persistent entrance- and exit-block | intra-procedural
  (per-pulmonary vein pair analysis and per-patient analysis
Safety events | periprocedural and 12 months
  Vascular access complications, pericardial effusion / tamponade, phrenic nerve paly (temporal or permanent), atrio-esophageal fistula, esophageal ulcer, pulmonary vein stenosis, systemic embolism, stroke, TIA, death, cardiovascular death

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic, University of Barcelona, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No